CLINICAL TRIAL: NCT03753256
Title: Evaluation of Optical Coherence Tomography in Dentistry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: Heidelberg Engineering GmbH (Industry)
Responsible Party: Principal Investigator, Sinan Sen, Senior Teaching and Research Assistant, University of Heidelberg Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: S-370/2015
Record Dates: First submitted 2016-04-20; First posted 2018-11-26 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Dental Caries; Tooth Demineralization
MeSH Terms: conditions — Dental Caries; Tooth Demineralization

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transbond XT (Active Comparator): Application of different orthodontic surface sealants to participants:
  Randomly assigned quadrants in this arm will receive a bonding primer (Transbond XT) The investigators will evaluate in this arm
  1. the development of demineralization
  2. its adverse effects after application
  Interventions: Device: Transbond XT
- Protecto®CaF2Nano (Experimental): Application of different orthodontic surface sealants to participants:
  Randomly assigned quadrants in this arm will receive an orthodontic surface sealant (Protecto®CaF2Nano).
  The investigators will evaluate in this arm
  1. its abrasion behavior and the development of demineralization
  2. its adverse effects after the application
  Interventions: Device: Protecto®CaF2Nano
- Pro Seal® (Experimental): Application of different orthodontic surface sealants to participants:
  Randomly assigned quadrants in this arm will receive an orthodontic surface sealant (Pro Seal®).
  The investigators will evaluate in this arm
  1. its abrasion behavior and the development of demineralization
  2. its adverse effects after the application
  Interventions: Device: Pro Seal®
- Opal® Seal (Experimental): Application of different orthodontic surface sealants to participants:
  Randomly assigned quadrants in this arm will receive an orthodontic surface sealant (Opal®Seal).
  The investigators will evaluate in this arm
  1. its abrasion behavior and the development of demineralization
  2. its adverse effects after the application
  Interventions: Device: Opal®Seal

INTERVENTIONS:
Device: Transbond XT — Application of
  • Transbond XT (activator comparator) to labial surfaces of teeth of randomized quadrants.
  Arms: Transbond XT
Device: Protecto®CaF2Nano — Application of
  • Protecto®CaF2Nano (orthodontic surface sealant) to labial surfaces of teeth of randomized quadrants.
  Arms: Protecto®CaF2Nano
Device: Pro Seal® — Application of
  • Protecto®CaF2Nano (orthodontic surface sealant) to labial surfaces of teeth of randomized quadrants.
  Arms: Pro Seal®
Device: Opal®Seal — Application of
  • Opal®Seal (orthodontic surface sealant) to labial surfaces of teeth of randomized quadrants.
  Arms: Opal® Seal

SUMMARY:
Optical coherence tomography (OCT) is a medical diagnostic tool, providing non-invasive, non-radiative and high resolution imaging. OCT has been established since many years in ophthalmology. In dentistry the diagnostic potential of OCT is currently increasingly being noticed. This clinical study includes two individual trials: (i) Longitudinal assessment of surface sealant thickness using optical coherence tomography and (ii) comparison of crevicular fluid levels of inflammatory cytokines after the application of surface sealants.

DETAILED DESCRIPTION:
Trial 1: Evaluation of the abrasion behavior of the orthodontic surface sealants Pro Seal®, Opal®Seal, and Protecto®CaF2Nano. The quadrants of 20 participants will be randomly assigned to four study groups. Using a split mouth design three commonly used orthodontic surface sealants (Pro Seal®, Opal®Seal, and Protecto®CaF2Nano) and a bonding primer (Transbond XT) which is used as a control will be applied to the labial surfaces of the teeth of the respective quadrants. The thickness changes of the orthodontic surface sealants and the development of enamel demineralization will be monitored at the day of the application and five additional time points (t1= 1 month, t2= 3 months, t3= 6 months, t4=9 months, t5= 12 months) using OCT.

Trial 2: Evaluation of Adverse effects of orthodontic surface sealants. 15 quadrants of the trial group described above (Trial1) will be randomly selected and gingival crevicular fluid (GCF) will be sampled in the respective quadrants at the day of bracket bonding prior (t0) and at three additional time points (t1= 30 min, t2= 60 min, t3= 90 min) after the application of surface sealants or the bonding primer, respectively. Analysis will be performed using magnetic Luminex screening assays for IL-8 (Interleukin 8), and IL-10 (Interleukin 10) and examined for inflammatory cytokines after the application of surface sealants.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic treatment need
* Informed consent from all patients and their parents or legal guardians after explaining of the study

Exclusion Criteria:

• withdrawn consent

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Abrasion behaviour of orthodontic surface sealants | The thickness changes of the orthodontic surface sealants and the development of enamel demineralization will be monitored at the day of the application and five additional time points (t1= 1 month, t2= 3 months, t3= 6 months, t4=9 months, t5= 12 months)
  Longitudinal assesment of surface sealant thickness using optical coherence tomography

SECONDARY OUTCOMES:
Adverse effects of orthodontic surface sealants | To assess cytokine levels GCF will be sampled at the day of bracket bonding prior (t0) and at three additional time points (t1= 30 min, t2= 60 min, t3= 90 min) after the application of surface sealants or the bonding primer, respectively.
  To evaluate possible adverse effects of orthodontic surface sealants in vivo gingival crevicular fluid will be sampled in the respective quadrants at the day of bracket bonding prior (t0) and at three additional time points (t1= 30 min, t2= 60 min, t3= 90 min) after the application of surface sealants or the bonding primer. Existing data on possible adverse effects of resin monomers from restorative composites or surface sealants were obtained using 3D tissue models; therefore, in the present study the investigators will attempt to evaluate possible adverse effects of commonly used smooth surface sealants on gingival tissues by analysing inflammatory cytokines in crevicular fluid of the participants after the application of surface sealants.To this end, the levels of the inflammatory cytokines (IL-8 (Interleukin 8), and IL-10 (Interleukin 10) in GCF will be assessed using multiplex analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Sen, Dr., Study Director — Department of Orthodontics and Dentofacial Orthopaedics, University of Heidelberg
Locations (1):
- Department of Orthodontics and Dentofacial Orthopaedics, University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alsayed EZ, Hariri I, Sadr A, Nakashima S, Bakhsh TA, Shimada Y, Sumi Y, Tagami J. Optical coherence tomography for evaluation of enamel and protective coatings. Dent Mater J. 2015;34(1):98-107. doi: 10.4012/dmj.2014-215. PMID 25748465
- [Result] Levin SM. Portasystemic shunts for portal hypertension: early and late results in a personal series of 140 operations. Vasc Surg. 1974 Jan-Feb;8(1):20-5. No abstract available. PMID 4544493
- [Result] Ryf S, Flury S, Palaniappan S, Lussi A, van Meerbeek B, Zimmerli B. Enamel loss and adhesive remnants following bracket removal and various clean-up procedures in vitro. Eur J Orthod. 2012 Feb;34(1):25-32. doi: 10.1093/ejo/cjq128. Epub 2011 Jan 12. PMID 21228118
- [Result] Lee SH, Lee JJ, Chung HJ, Park JT, Kim HJ. Dental optical coherence tomography: new potential diagnostic system for cracked-tooth syndrome. Surg Radiol Anat. 2016 Jan;38(1):49-54. doi: 10.1007/s00276-015-1514-8. Epub 2015 Jul 14. PMID 26168856
- [Result] Leao Filho JC, Braz AK, de Araujo RE, Tanaka OM, Pithon MM. Enamel Quality after Debonding: Evaluation by Optical Coherence Tomography. Braz Dent J. 2015 Jul-Aug;26(4):384-9. doi: 10.1590/0103-6440201300406. PMID 26312977
- [Result] Zingler S, Sommer A, Sen S, Saure D, Langer J, Guillon O, Lux CJ. Efficiency of powered systems for interproximal enamel reduction (IER) and enamel roughness before and after polishing-an in vitro study. Clin Oral Investig. 2016 Jun;20(5):933-42. doi: 10.1007/s00784-015-1585-2. Epub 2015 Sep 30. PMID 26419674
- [Derived] Sen S, Erber R, Orhan G, Zingler S, Lux CJ. OCT evaluation of orthodontic surface sealants: a 12-month follow-up randomized clinical trial. Clin Oral Investig. 2021 Mar;25(3):1547-1558. doi: 10.1007/s00784-020-03462-7. Epub 2020 Aug 13. PMID 32789656
- [Derived] Deurer N, Erber R, Orhan G, Zingler S, Lux CJ, Sen S. Abrasion of Pro Seal(R) and Opal(R) Seal by professional tooth cleaning protocols: results from an in vitro study and a randomized controlled trial. Eur J Orthod. 2020 Dec 2;42(6):596-604. doi: 10.1093/ejo/cjz096. PMID 31765473